CLINICAL TRIAL: NCT03931018
Title: Biomarkers of Acute Damage and Exposure/Consumption to Alcohol After an Experimental Administration of Alcohol Simulating a "Binge Drinking" Episode in Young Adults
Brief Title: Biomarkers of Alcohol After an Experimental Administration of Alcohol Simulating a "Binge Drinking" Episode
Acronym: BINGE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundació Institut Germans Trias i Pujol (Other)
Collaborators: Germans Trias i Pujol Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: HUGTP/BINGE/PNSD/1
Record Dates: First submitted 2019-02-08; First posted 2019-04-29 (Actual); Last update posted 2019-04-29 (Actual); Status verified 2019-04

CONDITIONS: Binge Drinking; Alcohol-Related Disorders
Keywords: "binge drinking"; "alcohol"; "pharmacokinetics"; "biomarkers"
MeSH Terms: conditions — Binge Drinking; Alcohol-Related Disorders | interventions — Ethanol

STUDY DESIGN:
Intervention Model Description: Two groups (one receiving 70 g and other receiving 100 g)
Who Masked: Participant
Masking Description: Simple Blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 70 grams alcohol (Experimental): Males and Females: Alcohol 70 grams (220 ml Vodka Absolut®), single dose, oral administration
  - 70 grams of alcohol mixed with zero orange soda without bubbles distributed in 6 glasses (total volume 900 ml) over a 2-hour period (20 minutes for glass)
  Interventions: Other: Alcohol
- 100 grams alcohol (Experimental): Males: Alcohol 100 grams (312 ml Vodka Absolut®), single dose, oral administration
  - 100 grams of alcohol mixed with zero orange soda without bubbles distributed in 6 glasses (total volume 900 ml) over a 2-hour period (20 minutes for glass)
  Interventions: Other: Alcohol

INTERVENTIONS:
Other: Alcohol — Administration of one dose of alcohol among two possible different doses (in males) or only one possible dose (in females) simulating a binge drinking episode under experimental conditions.

SUMMARY:
The purposes of this study are 1) to determine the pharmacokinetics of alcohol after experimental administration of alcohol simulating a "binge-drinking" episode in young adults 2) to determine the profile of biomarkers of acute damage and exposure/consumption to alcohol 3) to determine the pharmacokinetic parameters and evaluate the acute effects alcohol and its relationship with biomarkers.

DETAILED DESCRIPTION:
Binge drinking (BD) has become trendy among adolescents and young adults. It is defined as a pattern of drinking that reach blood alcohol concentration (BAC) to 80 mg/dl in a short period of time (2 hours), that typically occurs after 4 drinks for women and 5 drinks for men. Despite its high prevalence and association with morbidity and mortality, there are no previous experimental studies evaluating alcohol concentrations after a "binge drinking" episode neither its effects on biomarkers of acute damage and exposure/consumption.

The aims of this study are 1) to determine the pharmacokinetics of alcohol after experimental administration of alcohol simulating a "binge-drinking" episode in young adults 2) to determine the profile of biomarkers of acute damage and exposure/consumption to alcohol 3) to determine the pharmacokinetic parameters and evaluate the acute effects alcohol and its relationship with biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Understanding and accepting the study procedures and signing the informed consent.
* Male and females healthy volunteers (18-35 years old)
* Clinical history and physical examination demonstrating no organic or psychiatric disorders.
* The ECG and general blood and urine laboratory tests performed before the study should be within normal ranges. Minor or occasional changes from normal ranges are accepted if, in the investigator's opinion, considering the current state of the art, they are not clinically significant, are not life-threatening for the subjects and do not interfere with the product assessment. These changes and their non-relevance will be justified in writing specifically.
* Body weight between 60 and 85 kilograms for men and between 50 and 65 kg in for women. Lower or higher weights will be accepted, if the researchers considered that do not pose a risk to the subjects and do not interfere with the objectives of the study.
* BMI between 19-27 kg/m². Lower or higher BMIs will be allow, if the researchers considered that do not pose a risk to the subjects and do not interfere with the objectives of the study.
* Recreational use of alcohol at least 1 standard unit alcohol (standard drink)/day (accumulated in the week) and previous experiences in drunkenness and binge-drinking.
* Women with a regular menstrual cycle lasting between 26-32 days.

Exclusion Criteria:

* Not fill the inclusion criteria.
* History or clinical evidence of gastrointestinal, liver, renal or other disorders which may lead to suspecting a disorder in drug absorption, distribution, metabolism or excretion, or that suggest gastrointestinal irritation due to drugs.
* Present history of substance use disorder according to Diagnostic and Statistical Manual for Mental Disorders (DSM)-IV (except for nicotine). Past history of mild substance use disorder (corresponding to abuse substance according to DSM-IV) could be included.
* Blood donation 8 weeks before or participation in other clinical trials with drugs in the previous 12 weeks.
* Having suffered any organic disease or major surgery in the three months prior to the study start.
* Subjects with intolerance or serious adverse reactions to alcohol. Asian subjects with no intolerance or serious adverse reactions to alcohol could be included.
* Regular use of any drug in the month prior to the study sessions.The treatment with single or limited doses of symptomatic medicinal products in the week prior to the study sessions will not be a reason for exclusion if it is calculated that it has been cleared completely the day of the experimental session.
* Daily consumption >10 cigarettes.
* Daily consumption >20 grams of alcohol in women and >40 grams of alcohol in men.

Daily consumption >5 coffees, tea, cola refreshment or other stimulating drinks or containing xanthines in the three months prior to the study start.

* Subjects unable to understand the nature, consequences of the study and the procedures requested to be followed.
* Subjects with positive serology to Hepatitis B, C or HIV.
* Pregnant, breastfeeding women or those not use an method of contraception or not use an effective contraceptive (i.e. abstinence, intrauterine devices, barrier methods or partner vasectomy).

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
Area Under the Concentration-Time Curve (AUC 0-24h) of alcohol concentration in blood. | From pre-dose (baseline, 0 hours) to 0.33 hours (h), 0.66 h, 1.33 h, 1.66 h, 2 h, 2.33 h, 2.66 h, 3 h, 3.5 h, 4 h, 5 h, 6 h, 8 h, 10 h, 12 h and 24 h post-dose.
  Calculation of AUC of the concentrations of alcohol in blood.

SECONDARY OUTCOMES:
Area Under the Concentration-Time Curve (AUC 0-24h) of biomarkers of acute damage and exposure/consumption in blood. | From pre-dose (base-line, 0 hour), to 2.33 hour (h), 4 h, 6 h, 8 h, 24 h post-dose. Additional samples will be collected at 7,14 and 21 days post-administration
  Calculation of AUC of the concentrations of other biomarkers of exposure/consumption in blood.
Cumulative amount of biomarkers of exposure/consumption excreted into urine up to collection time of last measurable concentration. | From pre-dose (base-line, 0 hours (h)) and following intervals 0-2h, 2-4h, 4-6h, 6-8h, 8-10h, 10-12h and 12-24h to 24h post-administration
  Urine will be collected in intervals and the total amount of biomarkers of exposure/consumption will be calculated (ethylglucuronide and ethylsulfate)
Elimination half-life f the concentrations of alcohol in blood. | From pre-dose (baseline, 0 hours) to 0.33 h, 0.66 h, 1.33 h, 1.66 h, 2 h, 2.33 h, 2.66 h, 3 h, 3.5 h, 4 h, 5 h, 6 h, 8 h, 10 h, 12 h and 24 h post-dose
  Calculation of elimination half-life of the concentrations of alcohol in blood.
Area Under the Concentration-Time Curve (AUC 0-24h) of alcohol in breath (BrAC) | From pre-dose (baseline, 0 hours) to 0.33 h, 0.66 h, 1.33 h, 1.66 h, 2 h, 2.33 h, 2.66 h, 3 h, 3.5 h, 4 h, 5 h, 6 h, 8 h, 10 h, 12 h and 24 h post-dose
  Calculation of AUC of the concentrations of alcohol in breath (BrAC)
Change in blood pressure | From pre-dose (baseline, 0 hours) to 24 hours post-dose
  Blood pressure measured in mmHg
Change in heart rate | From pre-dose (baseline, 0 hours) to 24 hours post-dose
  Heart rate measured in beats per minute
Change in oral temperature | From pre-dose (baseline, 0 hours) to 24 hours post-dose
  Oral temperature measured in Celsius degrees
Change in drunkenness | From pre-dose (baseline, 0 hours) to 24 hours post-dose.
  Drunkenness will be measured using rate scales
Change in subjective effects | From pre-dose (baseline, 0 hours) to 24 hours post-dose.
  Subjective effects will be measured using rate scales
Number of Participants with Serious and Non-Serious Adverse Events | From pre-dose (baseline, 0 hours) to 21 days post-dose.
  Collection of adverse effects spontaneously reported by the participants and/or observed by the investigators.

CONTACTS AND LOCATIONS:
Overall Officials: Esther Papaseit, MD, PhD, Principal Investigator — Germans Trias i Pujol Hospital
Locations (1):
- Hospital Universitari Germans Trias i Pujol-Institut d'Investigació en Ciències de la Salut Germans Trias i Pujol (HUGTP-IGTP), Badalona, Barcelona, Spain